CLINICAL TRIAL: NCT06608212
Title: FIRST-2.5: Finerenone Research of Early Safety and Effectiveness, Part 2.5
Brief Title: An Observational Study to Learn More About How Safe Finerenone is and How Well it Works in People With Chronic Kidney Disease and Type 2 Diabetes in Routine Medical Care in the United States
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22663
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
Keywords: CKD; T2DM
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Finerenone group: Patients with chronic kidney disease (CKD) and type 2 diabetes (T2D) initiating finerenone. Retrospective analysis using secondary data collection from existing healthcare data from the US. Considered data sources include the HealthVerity Chronic Kidney Disease Masterset
  Interventions: Drug: Finerenone (Kerendia, BAY948862)
- Comparator group: Patients with chronic kidney disease (CKD) and type 2 diabetes (T2D) not using finerenone. Retrospective analysis using secondary data collection from existing healthcare data from the US. Considered data sources include the HealthVerity Chronic Kidney Disease Masterset
  Interventions: Drug: Others except finerenone

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY948862) — Follow clinical practice/administration.
  Groups: Finerenone group
Drug: Others except finerenone — Follow clinical practice/administration. The non-use finerenone treatment strategy will require individuals to be free of finerenone use.
  Groups: Comparator group

SUMMARY:
This is an observational study in which data from people with chronic kidney disease (CKD) and Type 2 diabetes mellitus (T2D) are collected and studied.

In observational studies, only observations are made without participants receiving any advice or any changes to healthcare.

CKD is a long-term condition in which the kidneys' ability to work properly gradually decreases over time. It is common in people with Type 2 diabetes mellitus (T2D), a condition in which glucose levels rise in the blood. People who have T2D and CKD may also develop heart disease over time.

The study drug, finerenone, is already approved for doctors to prescribe to people with CKD and T2D in the US. It blocks the activity of a protein involved in worsening kidney function.

The participants in this study are allowed to take finerenone as part of their regular care from their doctors.

The main purpose of the study is to learn about how safe finerenone is and how well it works in people with CKD and T2D in routine medical care. To do this, researchers will collect information about the time to first occurrence of any of the following heart-related problems for participants in the US who are taking finerenone and those who are not taking it:

* Heart attacks
* Hospitalization due to heart failure The data will come from the electronic healthcare records of people with CKD and T2D in the US who are allowed to take finerenone after July 2021.

Researchers will track participants' data and will follow them until the occurrence of heart-related problems, the participant's data is no longer available, there is a change in the participant's treatment strategy, or the end of the study.

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion criteria on or before Time 0 (Time 0 = finerenone initiation date) :

* Active registration or continuous enrolment for at least 365 days in the data source before Time 0 (days [-365, 0])
* No recorded use of finerenone before Time 0 (days [-all available, 0])
* Aged 18 years or older on Time 0
* Diagnosis of T2D at any time on or before Time 0 (days [-all available, 0])
* Having a diagnosis code indicating CKD stage 1, 2, 3, 4, or stage unspecified on or before Time 0 (days [-all available, 0])

Exclusion criteria on or before Time 0:

* Finerenone users who are hospitalized or admitted for an emergency department visit on Time 0
* Type 1 diabetes (T1D) at any time on or before Time
* Evidence of end-stage kidney disease (ESKD) at any time on or before Time 0
* A diagnosis of kidney cancer at any time on or before Time 0
* A diagnosis of adrenal insufficiency at any time on or before Time 0
* Evidence of hepatic impairment at any time on or before Time 0
* An eGFR measurement < 25 mL/min/1.73 m2 on or in the 90 days before Time 0
* Evidence of recent increased serum potassium or hyperkalaemia
* Use of a strong CYP3A4 inhibitor on or in the 183 days before Time 0
* Evidence of pregnancy measured on or in the 40 weeks before Time 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with CKD and T2D who are eligible for finerenone prescription after the approval of finerenone in the US. The study cohort will identify patients who initiate finerenone and a comparator group of individuals with CKD and T2D not using finerenone. All eligible adult individuals (aged ≥ 18 years) in the data source will be selected for the study cohort without sampling from the source population. There will be no restrictions of the study population based on sex, race, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of composite cardiovascular outcome | Retrospective analysis from July 2021 to June 2025
  The composite cardiovascular outcome includes an inpatient hospital diagnosis of fatal or nonfatal acute myocardial infarction or an inpatient hospitalisation with a primary diagnosis of heart failure.

SECONDARY OUTCOMES:
Time to the first occurrence of an inpatient hospital diagnosis of fatal or nonfatal acute myocardial infarction | Retrospective analysis from July 2021 to June 2025
Time to the first occurrence of an inpatient hospitalisation with a primary diagnosis of heart failure | Retrospective analysis from July 2021 to June 2025
Time to the first occurrence of an inpatient hospital or emergency department diagnosis of heart failure for participants without a history of heart failure | Retrospective analysis from July 2021 to June 2025
Time to occurrence of specific Urine Albumin-Creatine Ratio (UACR) decline thresholds | Retrospective analysis from July 2021 to June 2025
Time to the first occurrence of a hospitalisation or emergency department visit with a diagnosis code for hyperkalaemia | Retrospective analysis from July 2021 to June 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.